CLINICAL TRIAL: NCT01453907
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Dose, Dose-Escalation Study to Evaluate the Safety and Pharmacokinetics of ETI-204 in Healthy Subjects
Brief Title: Single Dose, Weight-Based, Dose-Escalation Study With Intravenous ETI-204 in Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Elusys Therapeutics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AH105
Record Dates: First submitted 2011-10-14; First posted 2011-10-18 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2011-10

CONDITIONS: Anthrax
MeSH Terms: conditions — Anthrax | interventions — obiltoxaximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ETI-204 (Experimental): ETI-204, Anthim
  Interventions: Drug: ETI-204, "Anthim"
- placebo (Sham Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ETI-204, "Anthim" — intravenously, single dose
  Other Names: ETI-204
  Arms: ETI-204
Drug: placebo — intravenously, single dose
  Arms: placebo

SUMMARY:
This study will determine the safety and PK of a single IV dose of ETI-204 in subjects 18 to 65 years of age. Three cohorts will be studied with subjects receiving ETI-204. This study will be randomized, double-blind and stratified by gender. Each cohort will contain 36 subjects (including at least four females), 30 who will receive ETI-204 and six who will receive placebo.

DETAILED DESCRIPTION:
Protocol AH-105 is a single center, randomized, double-blind, placebo-controlled, sequential, dose escalation study. It will evaluate the safety and PK of single IV doses of ETI-204 administered to approximately 108 healthy male and female subjects. At each dose level, 30 healthy subjects, including at least 4 females, will be randomly assigned to active drug, and at least 6 healthy subjects of both genders will be randomly assigned to matching placebo.

Description of Agent: ETI-204 is a monoclonal antibody (mAb) to protective antigen (PA) from Bacillus anthracis.

The study will consist of 3 phases: Screening, Inpatient, and Outpatient Follow-up. Enrollment criteria will be determined during the 21-day Screening Phase (Visit 1), following by a 3 night inpatient phase where eligible subjects will receive a single dose of IV ETI-204 or matching placebo as described above and undergo routine safety monitoring, dermatologic assessments, and blood draws at pre-specified time points. Subjects will be discharged from the center after collection of the 48-hour PK sample. During the subsequent 70-day outpatient follow-up phase, subjects will return to the center on Days 8, 15, 29, 43 and 71 for clinical laboratory testing (hematology and clinical chemistry), physical examinations and vital signs measurements, and routine safety monitoring. Blood samples for PK and anti-drug antibodies (ADA)will also be collected. The 70 day post-dosing follow-up in this study was selected to allow characterization for the PK profile of ETI-204 and the potential development of ADA.

ELIGIBILITY:
Inclusion Criteria: Subjects who meet all of the criteria shown below may be included in the study.

1. Healthy male or female subjects between 18 and 65 years of age.
2. Subjects with a body mass index (BMI) > 18.5 and < 35 kg/m2.
3. Female subjects of childbearing potential (not post-menopausal or surgically sterile) must have a negative urine β-hCG pregnancy test at Screening.
4. Female subjects of childbearing potential (not post-menopausal or surgically sterile) must use a medically accepted method of contraception for the duration of the study, including the 70-day follow-up period. Acceptable methods of contraception include abstinence, a barrier method with spermicide, an intrauterine device (IUD) or a hormonal contraceptive (oral, transdermal, implanted, or injected) in conjunction with a barrier method.
5. Male subjects must agree to practice abstinence or to use a condom with spermicide for the duration of the study, including the 70-day follow-up period.
6. The subject has no clinically significant abnormalities on the clinical laboratory tests (hematology, clinical chemistry, or urinalysis) or ECG at Screening.
7. Subject provides written informed consent.

Exclusion Criteria:Subjects who meet any of the criteria below will be excluded from participation in the study.

1. Subject requires regular use of a medication for a chronic condition.
2. Subject has a clinically significant comorbidity that would interfere with the completion of the study procedures or objectives, or would compromise the subject's safety.
3. Subject has a systolic blood pressure (BP) > 140 mm Hg or a diastolic BP > 90 mm Hg.
4. Subject has a systolic BP < 90 mm Hg.
5. Subject has current suspected drug or alcohol abuse as specified in the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) (American Psychiatric Association 2000).
6. Subject has a positive alcohol or drug test result at Screening and on Day -1
7. Subject has received an investigational agent within 30 days or 5 half-lives (whichever is longer) of Screening.
8. Subject has congenital or acquired immunodeficiency syndrome.
9. Subject has a positive test for Hepatitis B (surface antigen), Hepatitis C, or human immunodeficiency virus (HIV) at Screening.
10. Subject smokes > 3 cigarettes per day.
11. Subject has ever had prior treatment for anthrax exposure, prior anthrax infection, prior immunization with any anthrax vaccine or prior treatment with an investigational anthrax treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2011-10; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Primary Objective | 71 days
  To evaluate the safety of increasing doses of ETI-204 in healthy subjects

SECONDARY OUTCOMES:
Secondary Objective | 71 days
  To evaluate the PK of increasing singles doses of ETI-204 in healthy subjects.
  To evaluate the immunogenicity of ETI-204 following IV administration in healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor A Lisbon, M.D., M.P.H, Principal Investigator — Quintiles Phase One Services
Locations (1):
- Quintiles, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Nagy CF, Leach TS, Hoffman JH, Czech A, Carpenter SE, Guttendorf R. Pharmacokinetics and Tolerability of Obiltoxaximab: A Report of 5 Healthy Volunteer Studies. Clin Ther. 2016 Sep;38(9):2083-2097.e7. doi: 10.1016/j.clinthera.2016.07.170. Epub 2016 Aug 24. PMID 27568215